CLINICAL TRIAL: NCT04329351
Title: Impact of PTFE-d Barrier Intentionally Exposed in Guided Bone Regeneration to Ridge Preservation: Microbiological, Radiographic, Patient-centered Outcomes, Molecular Patter of Bone-related Markers and Implant Stabilization
Brief Title: Impact of PTFE-d Barrier Intentionally Exposed to Bucal Environment in Guided Bone Regeneration to Ridge Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fernanda Vieira Ribeiro (Other)
Responsible Party: Sponsor-Investigator, Fernanda Vieira Ribeiro, DDS, MS, PHD, Professor, Paulista University
Organization: Paulista University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBR-barrier exposed
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Ridge Preservation
Keywords: Alveolar Bone Loss; guided bone regeneration
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided bone regeneration Group (Experimental): After extraction, Guided bone regeneration was conducted using the PTFE-d membrane (CytoplastTM Ti-250 Titanium-Reinforced, Anterior Narrow 12 mm x 24 mm, Osteogenics, Lubbock, TX, USA) was customized with scissors and adjusted over the socket, exceeding three millimeters from its margins. Then, the membrane was inserted subperiostally under the buccal and palatal flaps with the help of the Molt detacher. Minimal flap reflection was performed to stabilize the membrane, which was maintained intentionally exposed to the oral environment. Before suturing, the passive stability of the membrane over the alveolus was confirmed, as well as the absence of folds or wrinkles in the membrane. The flaps were then be approached in the pre-extraction position and sutured with crossed sutures, aiming to increase the stability of the membrane, with PTFE 4-0 thread (Cytoplast PTFE, CS0618PREM, Osteogenics, Lubbock, TX, USA).
  Interventions: Procedure: Guided Bone regeneration
- Non-Guided bone regeneration group (Placebo Comparator): After extraction, no further treatment (No addition of Guided bone regeneration) was performed. The flaps were then repositioned and sutured with 5.0 nylon thread (Ethicon, Jonhson's Jonhson, São José dos Campos).
  Interventions: Procedure: Guided Bone regeneration

INTERVENTIONS:
Procedure: Guided Bone regeneration — Guided bone regeneration to ridge preservation

SUMMARY:
The aim of this clinical-laboratorial, paralel, randomized, prospective and controlled study was determine the impact of of PTFE-d barrier intentionally exposed to bucal environment in guided bone regeneration to ridge preservation, using microbiological, radiographic, patient-centered outcomes, molecular patter of bone-related markers and implant stabilization. Fourty individuals with tooth extraction indication and subsequent implant placement between upper pre-molars were recruited. Patients were randomly allocated in one of this groups, following tooth extraction: 1) GBR: sockets received GBR with d-PTFE membranes which was maintained intentionally exposed to bucal environment and removed after 28 days; and 2) Non-GBR: sockets did not receive additional therapy after extration. After 3 months, all patients received dental implants and temporary implant-supported prostheses. Patient-reported outcomes in terms of morbidity, swelling and interference with daily life were recorded at 3, 7, 14, 28, 35 and 42 days following dental extraction and in terms of esthetic outcomes after prosthesis instalation by using questionaries. Samples of biofilm at surface repair/barrier were obtained in both groups at 3 and 28 days after extraction (in the moment of barrier removal) to microbiological evaluation using Illumina HiSeq system. Computed tomography obtained imediatlly after extraction and before implant placement will be analised to evaluation of changes on ridge dimensions. After 3 months following extration, bone tissue biopsies will be harvested from the sites designed to receive dental implants to evaluation of imunoenzimatic pattern (DKK1, OPG, OC, OPN, TNF-α, SOST, RANKL, OSN e TRAP) and gene expression (TGF-β, BSP e COL-I) of bone-related markers using Luminex/Magpix and PCR Real-Time, respectivally. Afer imlpant placement, the implant stability quotient (ISQ) was determined. The results will be statistically compared after normality test, with the level of significance set at 5%.

DETAILED DESCRIPTION:
Study design This clinical-laboratorial, paralel, randomized, prospective and controlled study will be determine the impact of of PTFE-d barrier intentionally exposed to bucal environment in guided bone regeneration to ridge preservation, using microbiological, radiographic, patient-centered outcomes, molecular patter of bone-related markers and implant stabilization.

Experimental groups

Following local anesthesia, an intrasulcular incision was made around the tooth to be extracted and a mucoperiosteal flap was detached for adequate exposure of 3 mm of the alveolar crest adjacent to the alveolus. After, procedures for dislocation and dental removal were performed in a minimally invasive manner, using periotomes, levers and extractors, if necessary. Subsequently, irrigation with saline solution was performed and then, using specific software, patients will be randomly assigned to receive one of the following treatments:

GBR Group: After extraction, the PTFE-d membrane (CytoplastTM Ti-250 Titanium-Reinforced, Anterior Narrow 12 mm x 24 mm, Osteogenics, Lubbock, TX, USA) was customized with scissors and adjusted over the socket, exceeding three millimeters from its margins. Then, the membrane was inserted subperiostally under the buccal and palatal flaps with the help of the Molt detacher. Minimal flap reflection was performed to stabilize the membrane, which was maintained intentionally exposed to the oral environment. Before suturing, the passive stability of the membrane over the alveolus was confirmed, as well as the absence of folds or wrinkles in the membrane. The flaps were then be approached in the pre-extraction position and sutured with crossed sutures, aiming to increase the stability of the membrane, with PTFE 4-0 thread (Cytoplast PTFE, CS0618PREM, Osteogenics, Lubbock, TX, USA).

Non-GBR group: After extraction, no further treatment was performed. The flaps were then repositioned and sutured with 5.0 nylon thread (Ethicon, Jonhson's Jonhson, São José dos Campos).

Temporary adhesive prostheses adapted to adjacent teeth were installed and maintained until the moment of implant placement. The supragingival biofilm control was performed with mouthwashes of 0.12% chlorhexidine for a period of 4 weeks in all experimental groups. Pre-surgical anti-inflammatory therapy (dexamethasone 4 mg, single dose, 1 hour before the procedure) and postoperative analgesics (sodium dipyrone 500 mg, every 4 hours, for 3 days) were indicated. Patients were instructed to take analgesic medication only in case of pain during the period described above, being instructed to record the amount of medications ingested. Prophylactic systemic antimicrobial therapy was performed 1 hour before surgical procedures with 2 grams of Amoxicillin and the same medication will be prescribed for 7 days in the postoperative period, 500 mg every 8 hours.

Sutures were removed after 15 days. In the GBR group, the membrane was removed after the 28-day period, under anesthesia (Hoffmann et al. 2007, Carbonell et al. 2014, Cheon et al. 2017), being removed gently with the traction movement with the aid of a tweezers.

All patients were monitored monthly, throughout the study period, to observe periodontal maintenance and reinforce hygiene instructions.

Implants and Prostheses Placement Three months after the extraction, regardless of the experimental group, patients received dental implants. Therefore, they were molded for rehabilitation planning and surgical guides were made to be used in the implant placement surgery. In the surgical procedure, patients were submitted to local anesthesia and mucoperiosteal flaps were made for access and adequate exposure of the alveolar bone. After, drilling was performed to insert the implants. In both groups, single-stage implants were performed, with the immediate placement of provisional prostheses on implants. All surgeries were performed by the same operator (EKM).

After the experimental phase of the study, the definitive prostheses were installed. The sutures of the surgical procedures were performed with 5.0 nylon thread (Ethicon, Jonhson's Jonhson, São José dos Campos) and it was removed after 7 days. The supragingival biofilm control was performed with mouthwashes of 0.12% chlorhexidine for a period of 7 days after the surgery. Pre-surgical anti-inflammatory therapy (dexamethasone 4 mg, single dose, 1 hour before the procedure) and postoperative analgesics (sodium dipyrone 500 mg, every 4 hours, for 2 days) were indicated.

Clinical examination The same examiner (SB) performed all clinical measurements. To perform the intra-examiner calibration, 15 non-study individuals presenting dental implants were chosen. The examiner measured the peri-implant probing depth of all individuals twice within a 24-hour period. The intra-class correlation was calculated as 95% reproducibility.

Using a North Carolina/Colorvue probe (Hu-Friedy, Chicago, IL, USA), the following parameters were measured at four sites of the dental implants included in the study at baseline (before extration and GBR) and at 3-month follow-up: Probing Depth (PPD/mm), which was the distance from the bottom of the periodontal sulcus/pocket to the periodontal margin; Clinical Attachment Level (CAL/mm), which was the distance from the cement enamel junction to the bottom of the periodontal pocket.

Microbioma evaluation Microbiological assessments of the biofilm present on the barriers (GBR Group) and in the repair area (non-GBR Group) were made after 3 days of extraction and after 28 days (at the time of removal of the barrier in the GBR group).

The microbiological analysis will be done through the Sequencing Technique of the 16S gene by the Illumina HiSeq platform, which allows to determine the diversity and abundance of the microbial population in the same sample. This evaluation will be carried out at the Centralized Multi-User Laboratory of Functional Genomics.

Evaluation of parameters reported by the patient The assessment of patient-centered parameters concerning to symptoms related to morbidity and quality of life in the postoperative period will be carried out after 3, 7, 14, 28, 35 and 42 days of extraction, using questionnaires, based on a horizontal line of 100 mm (Visual Analog Scale; VAS).

Molecular evaluation of markers related to osteoclast / blastogenesis In the surgical procedure for placing dental implants, during the milling to prepare the bed, bone tissue will be removed using a disposable bone collector adapted to the vacuum pump / surgical aspirator. Part of the bone tissue sample will be used for analysis of gene expression and another part for immunoenzymatic analysis of different biomarkers related to osteoclast / blastogenesis. All molecular analyzes related to osteoclast / blastogenesis markers will be performed at the Dental Research Laboratory of the Headquarters Institution. All biopsies collected will be stored in a specific solution to avoid degradation of RNA (RNAlater®, Ambion Inc., Austin, TX).

Gene Expression Analysis RNA extraction: The removed tissues will be properly packed in a solution to avoid degradation of the RNA (RNAlater®, Ambion Inc., Austin, TX). The total RNA will be isolated by the TRIZOL reagent method (Gibco BRL, Life Technologies, Rockville, MD, USA). First, the RNAlater solution will be aspirated and the crushed sample will then be placed in the TRIZOL reagent, shaken for 30 seconds and incubated for 5 minutes at room temperature. After this period, chloroform (Sigma, St. Louis, MO, USA) will be added, stirred and centrifuged at 10,000 rpm for 15 minutes at a temperature of 4oC. The aqueous portion will be transferred to another tube to which isopropanol will be added, shaken, incubated for 20 minutes at a temperature of -20oC and centrifuged in the same way as described above. After this process, a pellet will be formed, which will be washed with chilled 75% ethanol and dried at room temperature. The RNA samples will be resuspended in approximately 50µl of water treated with diethylpyrocarbonate (DEPC) and stored at -70oC. The concentration of RNA will be determined using a spectrophotometer.

Treatment with DNAase will be performed and Real-time PCR (RT-PCR) will be conducted.Primers for GAPDH (reference gene), Transforming growth factor (TGF-β), Bone sialoprotein (BSP) and Collagen type I (COL-I) will be designed with the aid of a pGBRram developed specifically to design primers for LightCycler (Roche Diagnostics GmbH, Mannheim, Germany). All primers will be checked for specificity by checking the Melting curve using positive and negative controls. The reaction profile will be determined according to the formula suggested by the equipment manufacturer. For each of the "runs", water will be used as a negative control, and the product of the reactions will be quantified using the manufacturer's own pGBRram (LightCycler Relative Quantification Software - Roche Diagnostics GmbH). GAPDH will be used as the reference gene (housekeeping) for the normalization of values.

Immunoenzymatic Analysis Part of the bone tissue sample collected at the time of implant placement will be placed in sterile tubes containing 400μL of phosphate buffered saline (PBS) with 0.05% Tween-20. All samples will be stored at -20 ° C. Then, the tissue will be weighed, homogenized and dissolved in PBS to a final concentration of 100mg of tissue / mL. After stirring in Vortex for 10 minutes, each sample will be centrifuged at 370g for 5 minutes, the supernatant will be collected and stored at -70 ° C until use. To avoid protease activity, the entire procedure will be performed at 4 ° C. Dickkopf (DKK1), Sclerostin (SOST), Tumor necrosis factor (TNF-α), Osteoprotegerin (OPG), Osteocalcin (OC), Osteopontin (OPN) (HBNMAG-51K, Millipore Corporation, Billerica, MA, USA ), NF-κB binding activator receptor (RANKL) (HRNKLMAG-31K-01, Millipore Corporation, Billerica, MA, USA), Osteonectin (OSN) and Tartrate Resistant Acid Phosphatase (TRAP) (HCMBMAG-22K, Millipore Corporation, Billerica, MA, USA), will be determined using Luminex / MAGpix technology, which allows to determine the presence and to quantify in an absolute way the concentration of different markers in the same sample.

For this purpose, the analyzes will be performed in 96-well plates, with the help of the high-sensitivity panels mentioned above, following the manufacturer's instructions.The samples will be evaluated in duplicate and the average of the values obtained will be used to calculate the concentrations of each marker.

Tomographic Analysis CT scans of the patients will be obtained immediately after extraction and 3 months later (before implant placement). Tomographic examinations performed in the different periods will be analyzed for the rate of bone loss after extraction and preservation of the socket, both vertically and horizontally, through the Dental Slice software.

ELIGIBILITY:
Inclusion criteria:

* patients aged between 30 and 70 years old
* with a tooth indicated for extraction and subsequent rehabilitation with dental implant
* tooth extraction should be related to one of the teeth between maxillary premolars (premolar, canine, lateral or central incisor)
* the reasons for extraction may include the impossibility of restorations due to the presence of extensive caries lesions, prosthetic failures, root fractures or endodontic failures.
* the region to receive implants must present, radiographically, bone dimensions that allow the future placement of the dental implant and adequate prosthetic space for the subsequent prosthetic rehabilitation.
* at least three bone walls must be present at the time of extraction.

Exclusion criteria:

* pregnancy
* lactation
* current smoking or ex-smokers
* other systemic conditions that could affect bone metabolism (e.g., immunologic disorders)
* use of anti-inflammatory, bisphosphonate and immunosuppressive medications.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
tomographic changes in bone height | baseline and at 3-month
  tomographic changes in bone height

SECONDARY OUTCOMES:
Clinical attachament level | baseline and at 3-month
  Clinical Attachment Level (CAL/mm), which was the distance from the cement enamel junction to the bottom of the periodontal pocket
Probing Depth (PPD/mm) | baseline and at 3-month
  Probing Depth (PPD/mm), which was the distance from the bottom of the periodontal sulcus/pocket to the periodontal margin
Microbioma analysys | 3 days and 28 days
  Microbiological assessments of the biofilm present on the barriers (GBR Group) and in the repair area (non-GBR Group). The microbiological analysis will be done through the Sequencing Technique of the 16S gene by the Illumina HiSeq platform, which allows to determine the diversity and abundance of the microbial population in the same sample.
patient-centered parameters | 3, 7, 14, 28, 35 and 42 days
  The assessment of patient-centered parameters concerning to symptoms related to morbidity and quality of life in the postoperative period will be carried using questionnaires
Gene expression analysis of markers related to osteoclast / blastogenesis | 3 months
  In the surgical procedure for placing dental implants, during the milling to prepare the bed, bone tissue will be removed using a disposable bone collector adapted to the vacuum pump / surgical aspirator. Part of the bone tissue sample will be used for analysis of gene expression. Real Time PCR wil be performed to analyseTransforming growth factor (TGF-β), Bone sialoprotein (BSP) and Collagen type I (COL-I)
Imunoenzimatic analysis of markers related to osteoclast / blastogenesis | 3 months
  In the surgical procedure for placing dental implants, during the milling to prepare the bed, bone tissue will be removed using a disposable bone collector adapted to the vacuum pump / surgical aspirator. Part of the bone tissue sample will be used for analysis of molecules determined by Multipllex assay. Magpix/Lumimnex assay wil be performed to analyse Dickkopf (DKK1), Sclerostin (SOST), Tumor necrosis factor (TNF-α), Osteoprotegerin (OPG), Osteocalcin (OC), Osteopontin (OPN) (HBNMAG-51K, Millipore Corporation, Billerica, MA, USA ), NF-κB binding activator receptor (RANKL) (HRNKLMAG-31K-01, Millipore Corporation, Billerica, MA, USA), Osteonectin (OSN) and Tartrate Resistant Acid Phosphatase (TRAP) (HCMBMAG-22K, Millipore Corporation, Billerica, MA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Zaffalon Casati Marcio, Study Director — Paulista University
Locations (2):
- Brazil (2):
  - School of Dentistry - Paulista University UNIP, São Paulo, São Paulo
  - Fernanda Vieira Ribeiro, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braz SHG, Monteiro MF, Matumoto EK, Correa MG, Casarin RCV, Ribeiro FV, Cirano FR, Casati MZ, Pimentel SP. Microbial colonization in the partially exposed nonabsorbable membrane during alveolar ridge preservation. Clin Oral Investig. 2024 Jun 14;28(7):373. doi: 10.1007/s00784-024-05763-7. PMID 38874776
- [Derived] Matumoto EK, Correa MG, Couso-Queiruga E, Monteiro MF, Graham Z, Braz SHG, Ribeiro FV, Pimentel SP, Cirano FR, Casati MZ. Influence of partially exposed nonabsorbable membrane for alveolar ridge preservation: A randomized controlled trial. Clin Implant Dent Relat Res. 2023 Jun;25(3):447-457. doi: 10.1111/cid.13202. Epub 2023 Mar 22. PMID 36946359